CLINICAL TRIAL: NCT03927248
Title: Pilot Study of Nivolumab and Procaspase Activating Compound-1 (PAC-1) for
Brief Title: PAC-1 for Treatment of Refractory, Metastatic Kidney Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: funding issues
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REN-01
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab and PAC-1 (Experimental): Patient will be accrued and started on dose 1 level of PAC-1 (500 mg). If no DLT is observed in first cycle of therapy (28 days), dose of PAC-1 will be escalated to 625 mg in second cycle of therapy for the same patient. If patient remains on study and has no dose limiting toxicities, then in third cycle, dose will be escalated to 750 mg and continue in following cycles, if no dose adjustment is needed because of toxicities. Nivolumab will be administered by IV infusion at a dose of 480 mg.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — See description in Arms/Groups section
  Other Names: PAC-1

SUMMARY:
The primary objective of the pilot study is to determine activity of PAC-1 and nivolumab combination in subjects with metastatic renal cell carcinoma previously treated with immune checkpoint inhibitor therapy as assessed by objective response rate (ORR) using RECIST 1.1 criteria.

DETAILED DESCRIPTION:
PAC-1 in combination with nivolumab: The MTD will be determined using a modified-Fibonacci dose-escalation 3+3 design.

This pilot study will evaluate nivolumab in combination with PAC-1 in subjects with metastatic RCC. Nivolumab will be delivered by IV infusion on Day 1 and PAC-1 will be taken orally on Days 1-28 of each 28-day cycle, and response will be evaluated after every 2 cycles. Treatment will continue until disease progression (based on RECIST 1.1 criteria), unacceptable toxicity, subject refusal, or subject death either from progression of disease, the therapy itself, or from other causes. Subjects who voluntarily stop the study, have progressive disease, or unacceptable toxicities will be followed for survival every 3 months for 12 months from start of study medication

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Histologically or cytologically confirmed renal cell carcinoma.
3. Stage IV disease progressing on prior immune checkpoint inhibitor therapy
4. Patients must have Eastern Cooperative Oncology Group (ECOG) performance status 0-2 (Appendix 1).
5. Patients must have anticipated life expectancy greater than 3 months.
6. Patients must have measurable disease as defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20mm with conventional techniques or as ≥10mm with spiral CT scan by RECIST version 1.1 criteria. Baseline measurements and evaluation of all sites of disease must be obtained within 4 weeks prior to registration.
7. Palliative radiation must have been completed 2 weeks prior to the initiation of study therapy.
8. Patient with known brain metastases must have been treated at least 2 weeks prior to enrollment, be asymptomatic from brain metastases, stable on brain imaging, and not be receiving a supra-physiologic dose of steroids (>or = 10 mg prednisone daily or equivalent).
9. Women must not be pregnant and breast-feeding.

   * All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy.
   * Women of childbearing potential (WOCBP) must be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 6 months after the last dose of study medication. Patients of childbearing potential are those who have not been surgically sterilized or have not been free of menses > 1 year.
10. Male patients who are sexually active with WOCBP must agree to use an adequate method of contraception or abstain from sexual intercourse for at least one week prior to starting with the first dose of study therapy through 7 months after the last dose of study therapy.
11. Required Initial Laboratory Values (tested within 2 weeks prior to registration):

    * Leukocytes ≥2000/ μl
    * Hemoglobin >9.0 g/dL
    * Platelets ≥100,000/ μl
    * ANC ≥1,500/ μl
    * Serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula below):

      * Female CrCl = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL
      * Male CrCl = (140 - age in years) x weight in kg x 1.00
    * Total Bilirubin <1.5 mg/dl (except for subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dl)
    * SGOT (AST) <2.5 x ULN
    * ALP <2.5 x ULN in absence of liver metastases (<5 x ULN if liver metastases present
    * PTT <1.5 x ULN
12. The participant is capable of understanding and complying with the protocol and has signed informed consent document.

Exclusion Criteria

1. Active, known or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
2. Condition requiring systemic treatment with either corticosteroids (> or=10mg/day prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses >10 mg daily prednisone equivalents are permitted in the absence or active autoimmune disease.
3. Active hepatitis B or hepatitis C infection.
4. History of human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
5. New York Heart Association class III or IV congestive heart failure.
6. Corrected QT interval calculated by Fridericia formula (QTcF) > 500 ms within 14 days registration.
7. Cardiovascular disorders including unstable angina pectoris, clinically-significant cardiac arrhythmias, myocardial infarction or stroke (including transient ischemic attack [TIA], or other ischemic event) within 6 months prior to registration.
8. Active infection requiring intravenous systemic treatment.
9. History of organ transplant.
10. Inability to swallow intact tablets.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
To determine activity of PAC-1 and nivolumab | 12 months
  Assess by objective response rate (ORR) using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.

SECONDARY OUTCOMES:
to evaluate the safety profile of nivolumab in combination with PAC-1. | 12 months
  Toxicities will be defined according to NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
To measure 3- and 6-months progression-free survival (PFS) rate. | 12 months
  PFS will be determined by using RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hurley, MD, Principal Investigator — HealthPartners Institute